CLINICAL TRIAL: NCT06846086
Title: A Clinical Study to Assess the Cardioprotective Effects of Melatonin in Patients With Cardiomyopathy
Brief Title: Cardioprotective Effects of Melatonin in Patients With Cardiomyopathy
Acronym: CEMC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reem Alaa Abdel Samie, teacher assistant in faculty of pharmacy, delta university for science and technology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Melatonin cardioprotection
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cardiomyopathies
Keywords: cardiomyopathy; melatonin
MeSH Terms: conditions — Cardiomyopathies | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): patients will receive melatonin 10 mg once daily
  Interventions: Drug: Melatonin 10 MG
- Control group (Placebo Comparator): standard cardiomyopathy therapy for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 10 MG — Melatonin
  Arms: Interventional group
Drug: Placebo — placebo
  Arms: Control group

SUMMARY:
The aim of current study is to: Evaluate the cardioprotective effects of melatonin in patients with cardiomyopathy.

DETAILED DESCRIPTION:
Cardiomyopathy is a progressive and debilitating condition characterized by structural and functional abnormalities of the myocardium, often leading to impaired cardiac function, systemic congestion, and organ dysfunction. It affects millions of individuals worldwide, contributing significantly to morbidity and mortality despite advances in medical management. The pathophysiology of cardiomyopathy is complex and multifactorial, involving neurohormonal activation, oxidative stress, inflammation, and adverse cardiac remodeling. Standard treatments, such as angiotensin-converting enzyme (ACE) inhibitors, beta-blockers, and diuretics, have been shown to improve symptoms and slow disease progression; however, the prognosis remains poor for many patients, emphasizing the urgent need for novel therapeutic strategies.

Melatonin, a neurohormone primarily secreted by the pineal gland, has attracted considerable interest due to its diverse biological properties. Beyond its role in regulating circadian rhythms, melatonin exhibits potent antioxidant and anti-inflammatory effects. It scavenges free radicals, reduces lipid peroxidation, and modulates inflammatory pathways, thereby protecting mitochondrial function and cellular integrity. Experimental studies have demonstrated melatonin's ability to mitigate myocardial injury and improve cardiac function in animal models of cardiomyopathy. Preliminary clinical studies also suggest that melatonin supplementation may improve endothelial function, reduce sympathetic overactivity, and enhance overall cardiovascular health .

Mitochondrial dysfunction is a hallmark of cardiomyopathy. Melatonin has been shown to preserve mitochondrial function by maintaining mitochondrial membrane potential, preventing the opening of the mitochondrial permeability transition pore, and promoting mitophagy-the selective removal of damaged mitochondria. These actions help sustain ATP production and reduce cardiomyocyte apoptosis .

Melatonin's antioxidant capacity extends beyond direct scavenging; melatonin also upregulates the expression of antioxidant enzymes like superoxide dismutase (SOD), glutathione peroxidase (GPx), and catalase, while simultaneously inhibiting pro-oxidant enzymes. This dual mechanism makes it particularly effective in mitigating oxidative stress, a key contributor to the pathogenesis of numerous diseases, including cardiovascular disorders, neurodegenerative diseases like Alzheimer's and Parkinson's, diabetes, and cancer. In cardiovascular diseases, melatonin reduces lipid peroxidation and preserves mitochondrial function, protecting against ischemia-reperfusion injury. In neurodegenerative conditions, it minimizes neuronal oxidative damage and supports synaptic integrity. Furthermore, in diabetes, melatonin helps maintain pancreatic β-cell function by countering oxidative stress and inflammation. These multifaceted antioxidant properties make melatonin a promising therapeutic agent in oxidative stress-driven pathologies Given its safety profile and multifaceted mechanisms of action, melatonin holds promise as an adjunctive therapy in managing cardiomyopathy. Its ability to target oxidative stress, inflammation, and mitochondrial dysfunction addresses key pathological processes underlying the disease

In summary, melatonin exhibits several properties that may be beneficial in the context of cardiomyopathy. Ongoing research is essential to fully elucidate its therapeutic potential and to determine optimal dosing strategies for affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with a confirmed diagnosis of cardiomyopathy based on clinical, echocardiographic, or imaging findings. .
* Stable condition on standard cardiomyopathy medications (e.g., ACE inhibitors, beta-blockers).
* Ability to provide informed consent.

Exclusion Criteria:

* Recent hospitalization for cardiomyopathy exacerbation (within the last 3 months).
* Severe kidney or liver impairment.
* Use of other investigational drugs or antioxidants.
* Pregnancy or planning to be pregnant in the next 6 months
* Previous known hypersensitivity to melatonin.
* Presence of atrial fibrillation or other significant arrhythmias at baseline.
* Participation in another research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Measurement | baseline , up to 3 month
  Unit of Measure: mmHg (Systolic and Diastolic Blood Pressure).
  • Echocardiography.
Heart Rate (HR) Measurement | baseline, up to 3 month
  Unit of Measure: Beats per minute (bpm).
Echocardiographic Parameters | Baseline , up to 3 months.
  Parameters Measured:
  * Left Ventricular Ejection Fraction (LVEF) (%).
  * Left Ventricular End-Diastolic Diameter (LVEDD) (mm).
  * Left Ventricular End-Systolic Diameter (LVESD) (mm). GLS %
Echocardiographic Parameters | Baseline , up to 3 months.
  Parameters Measured:
  * Left Ventricular Ejection Fraction (LVEF) (%).
  * Left Ventricular End-Diastolic Diameter (LVEDD) (mm).
  * Left Ventricular End-Systolic Diameter (LVESD) (mm).
Serum Concentration of NT Pro- BNP | Baseline, up to 3 months.
  Changes in serum B-type Natriuretic Peptide (BNP) concentration from baseline to Week 12.

SECONDARY OUTCOMES:
composite clinical endpoint score | baseline , up to 3 month
  A composite score incorporating the following parameters:
  * All-cause mortality.
  * Hospitalization.
  * Quality of life (QoL) changes, assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
    • Scoring Details:
  * Scale Name: Kansas City Cardiomyopathy Questionnaire (KCCQ).
  * Score Range: 0-100.
  * Interpretation: Higher scores indicate better quality of life and clinical status, while lower scores indicate worse condition.
Biochemical Markers | baseline , up to 3 month
  * Cardiac biomarkers: Natriuretic peptides (e.g., BNP) for heart stress or damage.
  * Inflammatory markers: Interleukin-6 (IL-6) which may reflect systemic inflammation.
  * Antioxidant status: Malondialdehyde (MDA) using commerially available kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Dakahlia, Egypt, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: No